CLINICAL TRIAL: NCT01634945
Title: Aetiology, Prevention and Control of Anaemia in Sub-Saharan Africa - Work Package 2: Efficacy Study: Efficacy of 2 Iron Fortified Porridges and IPT for the Prevention of Anemia in Young Children in Côte d'Ivoire.
Brief Title: Efficacy of Iron Fortified Complementary Food and IPT of Malaria in Young Children in Côte d'Ivoire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IZ70Z0_123900/1
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Anemia
Keywords: anemia; malaria; malnutrition; iron fortification; intermittent preventive treatment; subsaharan africa; ivory coast; young children
MeSH Terms: conditions — Anemia; Malaria; Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- FeFum porridge + IPT of malaria (Experimental)
  Interventions: Drug: SP/Amodiaquine + FeFum fortified porridge
- IPT of malaria (Experimental)
  Interventions: Drug: SP/amodiaquine
- FeFum porridge (Experimental)
  Interventions: Dietary Supplement: FeFum fortified porridge
- FePP porridge (Experimental)
  Interventions: Dietary Supplement: Ferric pyrophosphate fortified porridge

INTERVENTIONS:
Drug: SP/amodiaquine — One dose of SP (500 mg sulfadoxine plus 25 mg pyrimethamine, or half of the dose if body weight =< 10 kg) and three daily doses of Amodiaquine (1. Day: 200 mg, 2. Day: 200 mg and 3. Day: 100 mg, or half of the dose each day if body weight =< 10 kg), every three months, i.e. 3 times during 9 consecutive months.
  Arms: IPT of malaria
Dietary Supplement: FeFum fortified porridge — 6 times per week supply of iron fortified porridge (25 g portion containing 5.8 mg of iron: 2 mg as NaFeEDTA + 3.8 mg as ferrous fumarate) for 9 months.
  Arms: FeFum porridge
Drug: SP/Amodiaquine + FeFum fortified porridge — One dose of SP (500 mg sulfadoxine plus 25 mg pyrimethamine, or half of the dose if body weight =< 10 kg) and three daily doses of Amodiaquine (1. Day: 200 mg, 2. Day: 200 mg and 3. Day: 100 mg, or half of the dose each day if body weight =< 10 kg), every three months, i.e. 3 times during 9 consecutive months.
  6 times per week supply of iron fortified porridge (25 g portion containing 5.8 mg of iron: 2 mg as NaFeEDTA + 3.8 mg as ferrous fumarate) for 9 months.
  Arms: FeFum porridge + IPT of malaria
Dietary Supplement: Ferric pyrophosphate fortified porridge — 6 days per week supply of iron fortified porridge (25 g portion containing 5.8 mg of iron: 2 mg as NaFeEDTA + 3.8 mg as ferric pyrophosphate) for 9 months.
  Arms: FePP porridge
Other: Placebo — Placebo of SP/Amodiaquine every 3 months for 9 months. No dietary intervention.
  Arms: Placebo

SUMMARY:
The proposed project is aimed at testing two interventions, namely a highly bioavailable iron compound and a combination of SP plus amodiaquine for intermittent preventive treatment (IPT) of malaria, to reduce anaemia in very young children.

DETAILED DESCRIPTION:
Efficacy study - ANAEMIA project Côte d'Ivoire The proposed project is aimed at testing two interventions, namely a highly bioavailable iron compound and a combination of SP plus amodiaquine for intermittent preventive treatment (IPT) of malaria, to reduce anaemia in very young children. The fortified product will be provided as porridge (Nutribon produced by PKL) with an optimized formula (2 mg in the form of NaFeEDTA and 3.8 mg in the form of ferrous fumarate) of the premix. In addition, we will assess the Nutribon product currently available on the market and we will compare it to an optimized premix formula. The current and the optimized formula contain each 2 mg iron in the form of NaFeEDTA. In addition to the NaFeEDTA the current premix contains 3.8 mg in the form of ferric pyrophosphate, which is less bioavailable than the 3.8 mg ferrous fumarate in the optimized formula. The study will be carried out between May and December 2012 which includes the rainy season (April - October) with its two peaks in Côte d'Ivoire and thus the period when malaria transmission is highest. The study will be implemented in a Health and Demographic Surveillance System in Taabo in Côte d'Ivoire and comprise 625 children between 12 to 36 months. 375 eligible infants will receive a fortified porridge (250 with the improved formula and 125 with the current formula), whereas 250 infants will continue with their local diet (control group). Infants receiving the optimized formula and infants in the control group will be randomly assigned to IPT of malaria (125 in each group) or placebo (125 in each group). Thus, infants can be assigned to one of the following five groups: 1. group (n=125): fortified porridge (optimized formula) and IPT of malaria 2. group (n=125): fortified porridge (optimized formula) and placebo 3. group (n=125): local diet and IPT of malaria and 4. group (n=125): local diet and placebo. 5. group (n=125): fortified porridge (current formula) and placebo, representing the current situation in Côte d'Ivoire in infants consuming fortified complementary food. This efficacy trial will deepen our understanding in preventing anaemia and the interaction of bioavailable iron compounds with an antimalarial drug and related conditions in very young children. Further, the study should demonstrate whether the earlier study failed to show an impact on anaemia due to the use of an iron compound that lacked bioavailability and/or using an antimalarial drug in the IPT intervention arm that lacked efficacy perhaps due to resistance by P. falciparum, or other yet to be investigated causes.

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 12 - 36 months, both sexes
* Absence of major systemic illnesses (as assessed by medical doctor upon initial full clinical assessment)
* Registered in DSS Taabo and anticipated residence in the study area for at least 1 year
* No severe anaemia, i.e. Hb ≥70 g/L in infants, as assessed by a Coulter Counter device
* No known or reported hypersensitivity to sulfadoxine-pyrimethamine, amodiaquine
* No known or reported history of significant chronic illness
* Written informed consent of parents or legal guardian

Exclusion Criteria:

* severe anaemia, i.e. Hb ≥70 g/L in infants, as assessed by a Coulter Counter device
* major systemic illnesses (as assessed by medical doctor upon initial full clinical assessment)
* known or reported hypersensitivity to albendazole, sulfadoxine-pyrimethamine, amodiaquine
* known or reported history of significant chronic illness

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 629 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | 9 months
  The study population will consist of 12 to 36-month-old infants in villages covered by the Taabo DSS site. Assuming a mean Hb of 97.3±19.6 g/l and that an increase of 8 g/l in Hb would be clinically relevant, and allowing for a dropout rate of 20%, we calculated that 125 infants per group were initially needed to achieve a power level of 90% at a 5% level of significance.

SECONDARY OUTCOMES:
Iron status indicators (SF, TfR) | 9 months
  The study population will consist of 12 to 36-month-old infants in villages covered by the Taabo DSS site.
Malaria prevalence | 9 months
  The study population will consist of 12 to 36-month-old infants in villages covered by the Taabo DSS site.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Wegmüller, Doctor, Principal Investigator — Swiss Federal Institute of Technology
Locations (1):
- Hopital General de Taabo Cite, Taabo Cite, Côte d’Ivoire

REFERENCES:
- [Derived] Glinz D, Wegmuller R, Ouattara M, Diakite VG, Aaron GJ, Hofer L, Zimmermann MB, Adiossan LG, Utzinger J, N'Goran EK, Hurrell RF. Iron Fortified Complementary Foods Containing a Mixture of Sodium Iron EDTA with Either Ferrous Fumarate or Ferric Pyrophosphate Reduce Iron Deficiency Anemia in 12- to 36-Month-Old Children in a Malaria Endemic Setting: A Secondary Analysis of a Cluster-Randomized Controlled Trial. Nutrients. 2017 Jul 14;9(7):759. doi: 10.3390/nu9070759. PMID 28708072
- [Derived] Glinz D, Hurrell RF, Ouattara M, Zimmermann MB, Brittenham GM, Adiossan LG, Righetti AA, Seifert B, Diakite VG, Utzinger J, N'Goran EK, Wegmuller R. The effect of iron-fortified complementary food and intermittent preventive treatment of malaria on anaemia in 12- to 36-month-old children: a cluster-randomised controlled trial. Malar J. 2015 Sep 17;14:347. doi: 10.1186/s12936-015-0872-3. PMID 26377199